CLINICAL TRIAL: NCT01515683
Title: Behavioral Support to Cancer Patients Before Anesthesia
Brief Title: Behavioral Support Before Anesthesia
Acronym: STØB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Marianne K. Thygesen, Development Nurse - Researcher, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AA
Record Dates: First submitted 2011-12-15; First posted 2012-01-24 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Nervousness; Life Experiences
Keywords: Nervousness before anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- An anaesthetic nurse (Experimental)
  Interventions: Behavioral: Only support from an anaesthetic nurse on the surgery ward
- Theatre nurse + An anaesthetic nurse (Active Comparator): Support from theatre nurse and an anaesthetic nurse
  Interventions: Behavioral: Support: a theatre nurse + an anaesthetic nurse
- A nurse from ward + an anaesthesic nurse (Experimental): Support from a nurse from the ward and an anaesthetic nurse
  Interventions: Behavioral: Support: a nurse from the ward + an anaesthetic nurse
- Optional relative + an anaesthetic nurse (Experimental): Support from an optional relative and an anaesthetic nurse
  Interventions: Behavioral: Optional relative supports

INTERVENTIONS:
Behavioral: Only support from an anaesthetic nurse on the surgery ward — Additional staff are only present if required by law.
  Other Names: Nursing care from an anaesthetic nurse
  Arms: An anaesthetic nurse
Behavioral: Support: a theatre nurse + an anaesthetic nurse — Theatre nurse stay with the patient, follow her to the operating table and stays with her until she is anaesthetized
  Other Names: Care from a theatre nurse
  Arms: Theatre nurse + An anaesthetic nurse
Behavioral: Support: a nurse from the ward + an anaesthetic nurse — A nurse from the ward follows the patient to the operating table and stays with her until she is anaesthetized.
  Other Names: Nursing care from a ward nurse
  Arms: A nurse from ward + an anaesthesic nurse
Behavioral: Optional relative supports — Optional relative follows the patient to the operating table and stays with her until she is anaesthetized
  Other Names: Care from an optional relative
  Arms: Optional relative + an anaesthetic nurse

SUMMARY:
Studies shows that reduced nervousness before anaesthesia may improve a course past anaesthesia. Therefore it is interesting to investigate how we can best help patients shortly before anaesthesia. A RCT with three intervention arms (with different personal support) and a control arm (with usual personal support) is therefore performed.

Hypothesis: Nervousness is reduced by the new interventions compared to the usual help provided.

DETAILED DESCRIPTION:
All patients receive behavioral support the last half hour before anaesthesia, but at different times and provided by persons with different connection to the patients.

The last two patients in all arms will be interviewed about their experiences with the help offered.

Statistic will provide results in the quantitative part of the study and analysis and interpretation following ideas of the French philosopher Poul Ricoeur will provide results in the qualitative part of the study.

ELIGIBILITY:
Inclusion Criteria:

* All Danish-speaking expected gynaecological cancer patients, who are offered open surgery at Odense University Hospital, who can speak for themselves and have the opportunity to have close relative to follow before anaesthesia and who accept participation.

Exclusion Criteria:

* Senility

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2008-12; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in nervousness at the operating table | Baseline and when the patient is on the operating table, on average 1½ days
  VAS score shown by patients and written down by the anesthetic nurse correcte to one decimal place.

SECONDARY OUTCOMES:
Satisfaction with help from healthcare professionals | A questionnaire at discharge, an expected average of three days
  A validated questionnaire is filed out by patients. The questionnaire have six items measuring satisfaction with help from healthcare professionals provided at the hospital.
Healthcare professional time spent | The last half an hour before anaesthesia
  Healthcare professional time spent on interventions: Healthcare professional time used with patient and relative half an hour before anaesthesia byond what is required by law

CONTACTS AND LOCATIONS:
Overall Officials: Ole Mogensen, Professor, Study Chair — Southern University of Denmark
Locations (1):
- Gynækologisk obstetrisk afdeling D, Odense Universitetshospital, Odense, Fyn, Denmark